CLINICAL TRIAL: NCT04239183
Title: BE1 Study Spain - CAPSULE SYSTEM FOR COLOSTOMATES
Acronym: BE1
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: B. Braun Medical SA (Industry)
Responsible Party: Sponsor
Other Study IDs: BE1
Record Dates: First submitted 2020-01-16; First posted 2020-01-23 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Quality of Life of Colostomized Patient
Keywords: stomy; stomatherapy; colestomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Stomatherapy — Demonstrate improvement of quality of life (difference of at least 5 points in the StomaQoL questionnaire (21)) among descending colostomy patients, establishing the following comparisons.

SUMMARY:
A comparative study on the improvement of quality of life of colostomized patients using the new Be1 device with capsule system.

DETAILED DESCRIPTION:
The primary objective is to demonstrate improvement of quality of life (difference of at least 5 points in the StomaQoL questionnaire) among descending colostomy patients, establishing the following comparisons:

1. Patients with recent surgery who after one month using a current two-piece mechanical device switch to the new Be1 device with capsule system versus patients who after one month continue to use the same current two-piece mechanical device during four months.
2. Patients who have been using a current two-piece mechanical device during more than 6 months after an ostomy and agree to switch to the new Be1 device with capsule system during four months.

The following secondary objectives have been defined:

* Assessment of patient satisfaction with the new Be1 device with capsule system versus a current two-piece mechanical device.
* Demonstration that the new Be1 device with capsule system improves the microbiota of the colostomized patient.

ELIGIBILITY:
Inclusion Criteria:

- Inclusion criteria groups 1 and 2

* Patients of at least 18 years of age.
* Recently operated patients with a descending colostomy.
* Patients with a non-retracted stoma measuring no more than 1.5 cm in height.
* Patients agreeing to participate in the study and who have signed the informed consent in accordance with the legal requirements.
* Patients who in the opinion of the stoma therapist are candidates for a two-piece mechanical device.

Inclusion criteria group 3

* Patients of at least 18 years of age.
* Patients with a descending colostomy for over 6 months and who carry a two-piece mechanical device.
* Patients with a non-retracted stoma measuring no more than 1.5 cm in height.
* Patients agreeing to participate in the study and who have signed the informed consent in accordance with the legal requirements
* Patients who in the opinion of the stoma therapist are candidates for use of the Be1 device with capsule system.

Exclusion Criteria:

Exclusion criteria groups 1 and 2

* Patients with cognitive impairment which in the opinion of the investigator would not allow completion of the questionnaire or could pose problems.
* Patients who are participating in another study.
* Patients with multiple stomas.
* Vulnerable patients or subjects under legal tutelage.
* Patients with known allergy to any of the components of the study product.
* Patients with a retracted stoma.
* Patients with a prolapsed stoma or a stoma measuring more than 1.5 cm in height.

Exclusion criteria group 3

* Patients with cognitive impairment which in the opinion of the investigator would not allow completion of the questionnaire or could pose problems.
* Patients who are participating in another study.
* Patients with multiple stomas.
* Vulnerable patients or subjects under legal tutelage.
* Patients with known allergy to any of the components of the study product.
* Patients with a retracted stoma.
* Patients with a prolapsed stoma or a stoma measuring more than 1.5 cm in height.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will involve descending colostomy patients. There are three study groups. Two of them will comprise new patients (recently subjected to surgery), while the third will consist of patients with an ostomy for at least 6 months (pre-existing patients).
  The sample size will comprise 240 patients (85 patients in the mentioned two groups and 70 in the third).
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2020-01 (Estimated); Primary Completion 2021-01 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
StomaQoL | 1 month
  to demonstrate improvement of quality of life (difference of at least 5 points in the StomaQoL questionnaire) among descending colostomy patients

SECONDARY OUTCOMES:
Questionnaire | 1 month
  Assessment of patient satisfaction with the new Be1 device with capsule system versus a current two-piece mechanical device.
Biota Analysis | 1 month
  Demonstration that the new Be1 device with capsule system improves the microbiota of the colostomized patient

IPD SHARING:
Plan to Share IPD: Undecided